CLINICAL TRIAL: NCT00143806
Title: Investigator-Initiated, Use Study of Alefacept (Amevive) in Combination With Tapering Doses of Cyclosporine in Patients With Moderate to Severe Psoriasis
Brief Title: Transitioning From Cyclosporine to Alefacept in Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Collaborators: Biogen (Industry)
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4513
Record Dates: First submitted 2005-08-31; First posted 2005-09-02 (Estimated); Last update posted 2009-01-05 (Estimated); Status verified 2008-12

CONDITIONS: Psoriasis
Keywords: psoriasis; cyclosporine; transition; alefacept
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Transitioning patients from cyclosporine to alefacept

SUMMARY:
The purpose of this study is to devise a safe and effective method for transitioning patients from cyclosporine to alefacept.

DETAILED DESCRIPTION:
The purpose of this study is to devise a safe and effective method for transitioning patients from cyclosporine to alefacept. Patients in the study are well controlled on cyclosporine and desire to switch to alefacept. The study is done in three phases. In Phase 1 (12 week duration) the two drugs will be overlapped, with cyclosporine slowly tapering. Both drugs will be discontinued after 12 weeks. In Phase 2 (12 weeks duration), patients are off both drugs. In Phase 3 (24 weeks long), patients are on a second course of alefacept alone for 12 weeks and then off for 12 weeks. Topical and UV light treatments are allowed throughout the study. Total length of study is one year.

ELIGIBILITY:
Inclusion Criteria

* Adult psoriasis patients (18 to 80 years old), who are well controlled on cyclosporine (Static PGA score of mild, minimal or clear) and who need or desire to stop cyclosporine and start alefacept.

Exclusion Criteria

* CD4 <400
* Active infection (other than trivial URI, etc.)
* History of AIDS or Hepatitis B, C
* Inability to understand consent or comply with study requirements
* Pregnancy or Lactation
* History of heart or liver disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13
Dates: Start 2003-10; Study Completion 2007-05

PRIMARY OUTCOMES:
Static physicians global assessment (PGA) and quality of life as measured by DLQI

CONTACTS AND LOCATIONS:
Overall Officials: Alice Gottlieb, MD, PhD, Principal Investigator — Rutgers, The State University of New Jersey
Locations (1):
- UMDNJ Clinical Research Center, New Brunswick, New Jersey, United States